CLINICAL TRIAL: NCT02274285
Title: Immunogenicity and Safety of the DTaP-IPV/Hib Vaccine SP0204) Given as Three-dose Primary and One-dose Booster Vaccinations Versus Co-administration of DTaP-IPV Vaccine (DD-687) and Hib Vaccine (DF-098) in Infants in Japan
Brief Title: DTaP-IPV/Hib Vaccine Primary & Booster Vaccinations Versus Co-administration of DTaP-IPV and Hib Vaccine in Japanese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: J2I02 (EFC13640); U1111-1143-9112 (Other: WHO)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Tetanus; Diphtheria; Pertussis; Poliomyelitis; Bacterial Meningitis
Keywords: Tetanus; Diphtheria; Pertussis; Poliomyelitis; Bacterial meningitis; DTaP-IPV/Hib Combination vaccine
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough; Poliomyelitis; Meningitis, Bacterial | interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (SP0204) (Experimental): Participants will receive DTaP-IPV/Hib vaccine administered subcutaneously
  Interventions: Biological: DTaP-IPV/Hib Combined vaccine
- Group B (control) (Active Comparator): Participants will be given a co-administration of DTaP-IPV vaccine and Hib vaccine subcutaneously
  Interventions: Biological: DTaP-IPV vaccine and Hib vaccine
- Group C (Experimental): Participants will receive DTaP-IPV/Hib vaccine administered intramuscularly
  Interventions: Biological: DTaP-IPV/Hib Combined vaccine

INTERVENTIONS:
Biological: DTaP-IPV/Hib Combined vaccine — 0.5 mL, Subcutaneously. 3 times, each given 3 to 8 weeks apart
  Other Names: SP0204
  Arms: Group A (SP0204)
Biological: DTaP-IPV vaccine and Hib vaccine — 0.5 mL each, Subcutaneously, 3 times, each given 3 to 8 weeks apart
  Other Names: DD 687; DF 098
  Arms: Group B (control)
Biological: DTaP-IPV/Hib Combined vaccine — 0.5 mL, Intramuscularly. 3 times, each given 4 to 8 weeks apart
  Other Names: SP0204
  Arms: Group C

SUMMARY:
Primary objective:

* To demonstrate the non-inferiority in terms of seroprotection rates (Hib antigen (PRP), Diphtheria, Tetanus, and Pertussis antigens (PT and FHA), and polio types 1, 2 and 3 antigens) of investigational arm (Group A: DTaP-IPV/Hib) versus control arm (Group B: DTaP-IPV and Hib vaccines administered at separate sites), one month after the primary vaccination (all antigens).

Secondary objectives:

* To describe immune responses against all vaccine antigens with no pre-specified hypothesis, and at all time points (pre-dose 1, post-dose 3, pre-dose 4 and post-dose 4) in the two study groups (Group A and Group B).
* To describe the safety after each dose of each vaccine in the two study groups (Group A and Group B).
* To describe immune responses against all vaccine antigens with no pre-specified hypothesis, and at all time points (pre-dose 1, post-dose 3, pre-dose 4 and post-dose 4 (Group C)

DETAILED DESCRIPTION:
Participants will be enrolled in two steps (Cohort 1 and Cohort 2). Step one will enroll Cohort 1 made of 40 participants randomized in two groups with a 1:1 ratio.

After review of the local and systemic adverse events occurring during the 7 Days following the first dose administered in these subjects, 2nd vaccination of Cohort 1 participants will resume and enrollment of the participants of Cohort number 2 will start. Step two will enroll Cohort 2 made of subjects randomized in two groups with a 1:1 ratio.

A sub-study Group C will be enrolled and will receive the vaccine by intramuscular route.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 months to 68 months inclusive (recommended 3 to 8 months for Groups A and B; 2 months for Group C) on the day of inclusion
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Fever ≥ 37.5°C (axillary temperature) on the day of inclusion
* Any serious disease whether acute or chronic
* Past or current medical history of Guillain-Barre syndrome, acute thrombocytopenic purpura or encephalopathy
* History of diphtheria, tetanus, pertussis, poliomyelitis and Haemophilus influenzae type b infections
* History of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* History of anaphylaxis to any of the study vaccine components
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis or Haemophilus influenzae type b infections with a trial vaccine or another vaccine
* Congenital or current acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Participation in another clinical trial preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Blood or blood-derived products received in the past or current or planned administration during the trial (including immunoglobulins)
* Any vaccination with live vaccines within the past 27 days preceding the first trial vaccination
* Any vaccination with inactivated vaccines within the past 6 days preceding the first trial vaccination
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or HIV infection
* Subject ineligible according to the Investigator's clinical judgment
* Identified as employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family member (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Ages: 2 Months to 68 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-05-28 (Actual); Study Completion 2016-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with anti-Diphtheria level ≥ 0.1 IU/mL post-dose 3 | 21 Days post-dose 3
  Anti-Diphtheria antibody titers will be assayed by neutralization test on Vero cells culture in comparison to the WHO equine antitoxin standard (seroneutralization)

SECONDARY OUTCOMES:
Percentage of participants with Seroprotection to vaccine antigens following vaccination | Day 0 (pre-vaccination ) and 21 Days post-dose 3
  Seroprotection is defined as: percentage of participants with anti-Diphtheria and anti Tetanus antibody levels ≥0.01, ≥0.1 and ≥1.0 IU/mL
Geometric Mean Titer (GMT) of antibodies to vaccine antigens following vaccination | 21 Days post-dose 3
  Anti-Diphtheria antibody titers will be assayed by neutralization test on Vero cells culture in comparison to the WHO equine antitoxin standard (seroneutralization)
Information concerning the safety in terms of solicited injection site and systemic reactions, unsolicited adverse events, and serious adverse events post vaccination with DTaP IPV/Hib vaccine. | Day 0 (post-vaccination) up to 21 days post each vaccination
  Solicited injection site reactions: Tenderness, Erythema, Swelling and Induration; Solicited Systemic Reactions: Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost and Irritability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi
Locations (12):
- Japan (12):
  - Aichi
  - Chiba
  - Fukui
  - Fukuoka
  - Gunma
  - Hokkaido
  - Miyagi
  - Nagano
  - Osaka
  - Shizuoka
  - Tokyo
  - Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Nakayama T, Vidor E, Tsuzuki D, Nishina S, Sasaki T, Ishii Y, Mizukami H, Tsuge H. Immunogenicity and safety of a DTaP-IPV/Hib pentavalent vaccine given as primary and booster vaccinations in healthy infants and toddlers in Japan. J Infect Chemother. 2020 Jul;26(7):651-659. doi: 10.1016/j.jiac.2019.11.012. Epub 2020 Apr 16. PMID 32307307